CLINICAL TRIAL: NCT06903676
Title: Utility of Trypsinogen -2 in Early Detection and Follow Up of Post-pancreatectomy Acute Pancreatitis (PPAP)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Nicholas J Zyromski, Professor of Surgery, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 25075
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Pancreatitis; Pancreatectomy
Keywords: Pancreatectomy; Post-pancreatectomy acute pancreatitis; PPAP
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Pancreatectomy Patients (Experimental): Patients who underwent pancreatectomy and are having their urine dipstick tested for Trypsinogen-2
  Interventions: Device: TRP-2 Urine Dipstick

INTERVENTIONS:
Device: TRP-2 Urine Dipstick — Urine dipstick testing for Trypsinogen-2

SUMMARY:
The goal of this study is to learn if urine trypsinogen can be used to diagnose post-pancreatectomy acute pancreatitis in patients undergoing pancreatectomy.

Participants will have their urine measured by dipsticks during and after their surgery.

DETAILED DESCRIPTION:
Patients will be identified utilizing preoperative scheduling and clinic visits. Patients undergoing any pancreatectomy (such as: pancreatoduodenectomy, distal pancreatectomy, duodenal preserving pancreatic head resection) will be identified. These patients will be educated about possible enrollment in the prospective study in the preoperative clinic or in the surgery preoperative area. If enrolled, these patients will receive the standard of care postoperative laboratory tests. These include, but are not limited to, postoperative serum amylase, drain amylase, complete blood counts, and complete or basic metabolic panels. These patients will have standard of care pathologic review of their operative specimens. These patients will also have their urine tested for TRP-2. This design will allow for the direct comparison of the TRP-2 dipstick tests against the standard of care serum amylase tests. Furthermore, the measuring of serum amylase will allow for the evaluation of post-pancreatectomy acute pancreatitis by the ISGPS definition.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years of age
* Undergoing elective pancreatectomy for any indication

Exclusion Criteria:

* Younger than 18 years of age
* Pregnant women
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Detection of PPAP by Urine Trypsinogen 2 | Day of surgery and post-operative days 1, 2 and 3
  TRP-2 will be measured in freshly obtained urine preoperatively as a control, intraoperatively at time of pancreas transection, in the post anesthesia recovery unit, and in the morning of POD 1-3. This will be measured by the Actim Pancreatitis urine dipstick test. This will be compared to standard of care serum amylase tests.

SECONDARY OUTCOMES:
Correlation of PPAP diagnosis | Postoperative Day 3
  PPAP diagnosis by Urine Trypsinogen 2 will be correlated with PPAP diagnosed by the International Study Group for Pancreatic Surgery (ISGPS) definition. PPAP, as defined by the ISGPS, requires (1) a sustained postoperative serum hyperamylasemia greater than the upper limit of normal for at least the first 48 hours postoperatively, (2) clinically relevant features, and (3) radiologic alterations consistent with PPAP.

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Health University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
This study is not planning to share IPD with other researchers. All IPD will be limited to secure encrypted servers by the institution. Only direct investigators for the study will have access to the IPD.